CLINICAL TRIAL: NCT07407920
Title: Optimization of Adjuvant Systemic Therapy in Patients With Early HER2-Positive (HER2+) Breast Cancer or Triple Negative Breast Cancer (TNBC) That Achieved a Pathological Complete Response (pCR) After Neoadjuvant Systemic Therapy and Do Not Have Molecular Residual Disease (MRD-Negative): A Phase II Clinical Trial (The MolecularPCR Trial)
Brief Title: Ph2 Study for Optimization of Adjunct Systemic Therapy in HER2+ Patients, MolecularPCR Trial
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2024-1206; NCI-2025-08252 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 2024-1206 (Other: M D Anderson Cancer Center); P30CA016672 (NIH)
Record Dates: First submitted 2026-02-06; First posted 2026-02-12 (Actual); Last update posted 2026-02-12 (Actual); Status verified 2026-02

CONDITIONS: Anatomic Stage I Breast Cancer AJCC v8; Anatomic Stage II Breast Cancer AJCC v8; Early Stage HER2-Positive Breast Carcinoma; Early Stage Triple-Negative Breast Carcinoma
MeSH Terms: interventions — Specimen Handling; Steroids; Hormones; pembrolizumab; pertuzumab; 2C4 antibody; Trastuzumab; CT-P6; PF-05280014; trastuzumab biosimilar HLX02; Ogivri; Ontruzant

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- Cohort 1 (Triple negative breast cancer) (Experimental): Patients may receive 1 to 3 cycles of standard of care treatment with pembrolizumab. Patients with a positive ctDNA test 4-6 weeks after surgery continue to receive standard of care treatment per their treating physician in the absence of disease progression or unacceptable toxicity. Patients with a negative ctDNA test will not receive further treatment with pembrolizumab and will undergo monitoring with ctDNA tests every 3 months for 3 years in the absence of disease progression. Patients undergo blood sample collection throughout the study.
  Interventions: Procedure: Biospecimen Collection; Biological: Pembrolizumab
- Cohort 2 (HER2 positive breast cancer) (Experimental): Patients may receive 1 to 3 cycles of standard of care treatment with trastuzumab with or without pertuzumab. Patients with a positive ctDNA test 4-6 weeks after surgery continue to receive standard of care treatment per their treating physician in the absence of disease progression or unacceptable toxicity. Patients with a negative ctDNA test will not receive further treatment with pembrolizumab and will undergo monitoring with ctDNA tests every 3 months for 3 years in the absence of disease progression. Patients may receive standard of care endocrine therapy per their treating physician throughout the study. Patients undergo blood sample collection throughout the study.
  Interventions: Procedure: Biospecimen Collection; Drug: Hormone Therapy; Biological: Pertuzumab; Biological: Trastuzumab

INTERVENTIONS:
Procedure: Biospecimen Collection — Undergo blood sample collection
  Other Names: Biological Sample Collection; Biospecimen Collected; Specimen Collection
Drug: Hormone Therapy — Given standard of care endocrine therapy
  Other Names: Chemotherapy-Hormones/Steroids; Endocrine Therapy; Hormonal; Hormonal Therapy; Hormonal Treatment; hormone treatment; Hormones
  Arms: Cohort 2 (HER2 positive breast cancer)
Biological: Pembrolizumab — Given pembrolizumab
  Other Names: BCD-201; GME 751; GME751; Keytruda; Lambrolizumab; MK 3475; MK-3475; MK3475; Pembrolizumab Biosimilar BCD-201; Pembrolizumab Biosimilar GME751; Pembrolizumab Biosimilar QL2107; Pembrolizumab Biosimilar RPH-075; Pembrolizumab Biosimilar SB27; QL2107; RPH 075; RPH-075; RPH075; SB 27; SB-27; SB27; SCH 900475; SCH-900475; SCH900475
  Arms: Cohort 1 (Triple negative breast cancer)
Biological: Pertuzumab — Given pertuzumab
  Other Names: 2C4; 2C4 Antibody; BCD-178; EG1206A; HLX11; HS627; MoAb 2C4; Monoclonal Antibody 2C4; Omnitarg; Perjeta; Pertuzumab Biosimilar BCD-178; Pertuzumab Biosimilar EG1206A; Pertuzumab Biosimilar HLX11; Pertuzumab Biosimilar HS627; Pertuzumab Biosimilar TQB2440; Pertuzumab-dpzb; Poherdy; Rhumab 2C4; rhuMAb2C4; RO4368451; TQB 2440; TQB-2440; TQB2440
  Arms: Cohort 2 (HER2 positive breast cancer)
Biological: Trastuzumab — Given trastuzumab
  Other Names: ABP 980; ALT02; Biceltis; CANMab; CT-P06; CT-P6; Herceptin; Herceptin Biosimilar PF-05280014; Herceptin Trastuzumab Biosimilar PF-05280014; Hercessi; Herclon; Hertraz; Herwenda; Herzuma; HLX 02; HLX-02; HLX02; Kanjinti; Ogivri; Ontruzant; PF 05280014; PF-05280014; PF05280014; QL 1701; QL-1701; QL1701; rhuMAb HER2; RO0452317; SB3; Trastuzumab Biosimilar ABP 980; Trastuzumab Biosimilar ALT02; Trastuzumab Biosimilar CT-P6; trastuzumab biosimilar EG12014; Trastuzumab Biosimilar HLX02; Trastuzumab Biosimilar PF-05280014; Trastuzumab Biosimilar QL1701; Trastuzumab Biosimilar SB3; Trastuzumab Biosimilar SIBP-01; Trastuzumab-anns; Trastuzumab-dkst; Trastuzumab-dttb; Trastuzumab-herw; Trastuzumab-pkrb; Trastuzumab-qyyp; Trastuzumab-strf; Trastuzumab-zerc; Trazimera; Zercepac
  Arms: Cohort 2 (HER2 positive breast cancer)

SUMMARY:
This phase II trial tests reduced post surgery (adjuvant) therapy for patients with early breast cancer who have confirmed that the disease has responded completely (pathologic complete response) after pre surgical treatment (neoadjuvant) therapy and do not have any tumor genetic material (molecular residual disease) circulating in their blood. Standard of care treatment after surgery consists of 1 year of pembrolizumab for patients with triple negative breast cancer or trastuzumab with or without pertuzumab to complete 1 year of treatment. Immunotherapy with monoclonal antibodies, such as pembrolizumab, may help the body's immune system attack the cancer, and may interfere with the ability of tumor cells to grow and spread. Pertuzumab and trastuzumab are monoclonal antibodies and forms of targeted therapy that attach to a receptor protein called HER2. HER2 is found on some cancer cells. When pertuzumab or trastuzumab attach to HER2, the signals that tell the cells to grow are blocked and the tumor cell may be marked for destruction by the body's immune system. Lowering the total amount of cancer therapy after breast surgery, may continue to keep the great tumor response to treatment, and may help lower the amount of side effects patients have.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To determine the 3-year event free survival (EFS) after breast surgery in patients with early triple negative breast cancer (TNBC) that achieve a pathologic complete response (pCR) after neoadjuvant systemic therapy (NST) with a pembrolizumab plus chemotherapy-based regimen and are minimal residual disease (MRD)-negative (negative circulating tumor deoxyribonucleic acid [ctDNA] with the NeXT Personal™ assay) at 4-6 weeks after breast surgery and discontinue standard of care (SOC) adjuvant pembrolizumab.

II. To determine the 3-year EFS after breast surgery in patients with early HER2+ breast cancer that achieve a pCR after NST with a trastuzumab and pertuzumab plus chemotherapy-based regimen and are MRD-negative (negative ctDNA with the NeXT Personal™ assay) at 4-6 weeks after breast surgery and discontinue SOC adjuvant trastuzumab and pertuzumab.

SECONDARY OBJECTIVES:

I. To estimate the rate of conversion from negative to positive ctDNA and time to conversion from negative to positive ctDNA among patients who undergo de-escalation of SOC adjuvant systemic therapy.

II. To establish the prevalence of patients with early TNBC or early HER2+ breast cancer who achieve a pCR after receiving NST and have a positive ctDNA with the NeXT Personal™ assay at 4-6 weeks after breast surgery.

III. To determine the 3-year EFS after breast surgery in patients with early HER2+ breast cancer or early TNBC that achieve a pCR after NST and have a positive ctDNA with the NeXT Personal™ assay at 4-6 weeks after breast surgery.

OUTLINE: Patients with triple negative breast cancer are assigned to cohort 1, patients with HER2 positive breast cancer are assigned to cohort 2.

COHORT 1: Patients may receive 1 to 3 cycles of standard of care treatment with pembrolizumab. Patients with a positive ctDNA test 4-6 weeks after surgery continue to receive standard of care treatment per their treating physician in the absence of disease progression or unacceptable toxicity. Patients with a negative ctDNA test will not receive further treatment with pembrolizumab and will undergo monitoring with ctDNA tests every 3 months for 3 years in the absence of disease progression.

COHORT 2: Patients may receive 1 to 3 cycles of standard of care treatment with trastuzumab with or without pertuzumab. Patients with a positive ctDNA test 4-6 weeks after surgery continue to receive standard of care treatment per their treating physician in the absence of disease progression or unacceptable toxicity. Patients with a negative ctDNA test will not receive further treatment with pembrolizumab and will undergo monitoring with ctDNA tests every 3 months for 3 years in the absence of disease progression. Patients may receive standard of care endocrine therapy per their treating physician throughout the study.

ELIGIBILITY:
Inclusion Criteria:

* EARLY HER2 POSITIVE (+) BREAST CANCER COHORT: Female or male with a diagnosis of biopsy proven invasive breast cancer HER2+, hormone (estrogen and progesterone)-receptor positive or negative. The HER2 status (following American Society of Clinical Oncology [ASCO]/College of American Pathologists [CAP] guidelines) and hormone-receptor status will be determined according to institutional (local) guidelines
* EARLY TNBC COHORT: Female or male with a diagnosis of biopsy proven invasive TNBC (estrogen and progesterone receptor < 10%). The HER2 status (following ASCO/CAP guidelines) and hormone-receptor status will be determined according to institutional (local) guidelines
* FOR BOTH HER2+ AND TNBC COHORTS: Invasive breast cancer of any tumor histologic grade and/or nuclear grade, and any tumor histological subtype including but not limited to infiltrating ductal carcinoma, infiltrating lobular carcinoma, mucinous carcinoma, papillary carcinoma, tubular carcinoma, metaplastic carcinoma, and mixed histology
* FOR BOTH HER2+ AND TNBC COHORTS: Clinical tumor stage (per American Joint Committee on Cancer [AJCC] 8th edition): T1-4, N0-2a, M0. Patients who have a diagnosis of inflammatory breast cancer are eligible. Patients should not have clinical evidence of locoregional or distant metastatic breast cancer
* EARLY HER2+ BREAST CANCER COHORT: Have completed NST with a trastuzumab plus pertuzumab and chemotherapy-based regimen (for example, docetaxel plus minus carboplatin plus trastuzumab plus pertuzumab known as the docetaxel/pertuzumab/trastuzumab [THP]/carboplatin/paclitaxel/pertuzumab/trastuzumab [TCHP] regimens) followed by definitive breast surgery where the surgical pathology reports a pCR (ypT0-Tis, ypN0) and are willing to discontinue adjuvant trastuzumab plus pertuzumab
* EARLY TNBC COHORT: Have completed NST with a pembrolizumab plus chemotherapy-based regimen (for example, the KEYNOTE-522 regimen which is paclitaxel plus carboplatin plus pembrolizumab followed by doxorubicin plus cyclophosphamide plus pembrolizumab) followed by definitive breast surgery where the surgical pathology reports a pCR (ypT0-Tis, ypN0) and are willing to discontinue adjuvant pembrolizumab
* The surgical pathology report needs to show a pCR (ypT0-Tis, ypN0) for a patient to be able to participate in this study and all enrolled patients should be willing to discontinue standard adjuvant systemic therapy
* FOR BOTH HER2+ AND TNBC COHORTS: Adequate archival tumor tissue from the core diagnostic biopsy (per Personalis)
* FOR BOTH HER2+ AND TNBC COHORTS: Age ≥ 18 years
* FOR BOTH HER2+ AND TNBC COHORTS: Eastern Cooperative Oncology Group (ECOG) performance status ≤ 2 (Karnofsky ≥ 60%)
* FOR BOTH HER2+ AND TNBC COHORTS: Absolute neutrophil count ≥ 1,000/mcL
* FOR BOTH HER2+ AND TNBC COHORTS: Hemoglobin ≥ 9.0 g/dL
* FOR BOTH HER2+ AND TNBC COHORTS: Platelets ≥ 100,000/mcL
* FOR BOTH HER2+ AND TNBC COHORTS: Total bilirubin ≤ 1.5 institutional upper limit of normal (ULN); patients with Gilbert's syndrome (if direct bilirubin <1.5 x institutional ULN)
* FOR BOTH HER2+ AND TNBC COHORTS: Aspartate aminotransferase (AST)(serum glutamic oxaloacetic transaminase [SGOT])/ alanine aminotransferase (ALT) (serum glutamic pyruvic transaminase [SGPT]) ≤ 3 × institutional ULN
* FOR BOTH HER2+ AND TNBC COHORTS: Creatinine ≤ 1.5 mg/dL
* FOR BOTH HER2+ AND TNBC COHORTS: For patients with evidence of chronic hepatitis B virus (HBV) infection, the HBV viral load must be undetectable on suppressive therapy, if indicated
* FOR BOTH HER2+ AND TNBC COHORTS: Patients with a history of hepatitis C virus (HCV) infection must have been treated and cured. For patients with HCV infection who are currently on treatment, they are eligible if they have an undetectable HCV viral load
* FOR BOTH HER2+ AND TNBC COHORTS: Human immunodeficiency virus (HIV)-infected patients on effective anti-retroviral therapy with undetectable viral load within 6 months are eligible
* FOR BOTH HER2+ AND TNBC COHORTS: Pre- and postmenopausal women are eligible
* FOR BOTH HER2+ AND TNBC COHORTS: Ability to understand and the willingness to sign a written informed consent document

Exclusion Criteria:

* Patients with tumor stage of cN2b or cN3 are not eligible
* History of other malignancies besides breast cancer within the past 5 years, except cervical cancer in situ, melanoma in situ, basal cell carcinoma of the skin, or squamous cell carcinoma of the skin
* Patients who are receiving any other anti-cancer investigational agents
* Patients with known cancer metastases from any site
* Patients with uncontrolled intercurrent illness including but not limited to active infection, symptomatic congestive heart failure, unstable angina pectoris, symptomatic cardiac arrythmias
* Patients with psychiatric illness/social situations that would limit compliance with study requirements
* Blood transfusion within 2 weeks before collection of blood for ctDNA testing
* Patients who have received 4 or more cycles of SOC adjuvant trastuzumab/pertuzumab (HER2+) or 4 or more cycles of SOC adjuvant pembrolizumab (TNBC)
* Pregnant women are not eligible to participate in this study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2025-10-09 (Actual); Primary Completion 2026-09-30 (Estimated); Study Completion 2027-09-30 (Estimated)

PRIMARY OUTCOMES:
Event free survival (EFS) | From breast surgery to evidence of clinical locoregional or distant recurrence of breast cancer or death from breast cancer, up to 3 years
  Will be independently estimated for each cohort, along with corresponding 95% confidence intervals using Kaplan-Meier method.

SECONDARY OUTCOMES:
Rate of conversion from negative to positive circulating tumor deoxyribonucleic acid (ctDNA) | Up to 3 years
  95% confidence interval will be calculated by cohort using the Clopper-Pearson method.
Time to conversion from negative to positive ctDNA | Up to 3 years
  Will be estimated using the Kaplan-Meier method.
Prevalence of patients with pathologic complete response (pCR) rate after receiving neoadjuvant systemic therapy (NST) and have positive ctDNA | At 4-6 weeks after breast surgery
  The 95% confidence intervals for the prevalence estimates will be calculated using Clopper-Pearson method.
EFS in patients that achieve pCR after NST and have a positive ctDNA | From breast surgery to evidence of clinical locoregional or distant recurrence of breast cancer or death from breast cancer, up to 3 years
  EFS at 3 years with their 95% confidence intervals will be estimated using Kaplan-Meier method. Log-rank test will be performed to test the difference in time-to-event distributions between patient groups.

CONTACTS AND LOCATIONS:
Overall Officials: Vicente Valero, MD, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- M D Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: MD Anderson Cancer Center — http://www.mdanderson.org